CLINICAL TRIAL: NCT02508051
Title: Make a Journal Feel as if it Was Mailed Back From the Future Rather Than the Past so the Reader Will be More Likely to Read and Retain Journal Content
Brief Title: Make a Journal Feel as if it Was Mailed Back From the Future
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never received funding
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1506016077
Record Dates: First submitted 2015-07-23; First posted 2015-07-24 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Knowledge Bases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No daily emails (No Intervention): The usual care group will receive no intervention except for a reminder every six months to take a test of journal-based CME questions from 2 anesthesiology journals
- Article email links (Placebo Comparator): The email link group will get e-mailed web links to different specific articles, including articles on which the CME questions are based, published in 2 anesthesiology journals Monday through Friday with a reminder to take the same test every six months
  Interventions: Behavioral: Article email links
- Blog email links (Experimental): The experimental group will get e-mailed web links to blogs Monday through Friday based on the same specific articles as in group 2; each daily blog will focus on a specific article, including articles on which CME questions are based, the blogs will have web links to the articles on which they are based and every six months group 3 will get a reminder to take the same test.
  Interventions: Behavioral: Blog email links

INTERVENTIONS:
Behavioral: Article email links — Email links to specific articles, published in 2 journals M-Fr with a reminder to take the same test every six month
  Arms: Article email links
Behavioral: Blog email links — Emailed web links to blog posts M-Fr based on the same articles as in Email links group; each blog post will focus on a specific article with links to the corresponding article. Every six months group 3 will get a reminder to take the same test.
  Arms: Blog email links

SUMMARY:
Optimal patient care hinges on physicians remaining up to date with developing medical knowledge. With ever increasing clinical demands however, the ability of physicians to do this is compromised. While the structure of journal based reports requires the devotion of significant time to glean emerging medical findings, social media can grab an individual's attention and then direct them to external media sites, so as to obtain more specific and detailed information of emerging medical findings. If medical journals were to fully embrace social media, physicians would have a more time-cost effective means for staying up to date.

Specific aims Using the investigator's experience as editors of two medical education based blogs, the Specific Aims of this project is to determine if a combined journal and social media-based education strategy will be more likely to continuously engage physicians. The investigators will specifically test whether physicians who access a medical journal blog will have better knowledge of the information contained in a journal, measured by CME-based questions of journal articles than they would if they only received links to the journal's site.

Specifically, the investigators will randomize participants into 3 groups with all interventions done by e-mail: group 1 is the usual care group, and will receive no intervention except for a reminder every six months to take a test of journal-based Continuing Medical Education (CME) questions from 2 anesthesiology journals; group 2 will get e-mailed web links to different specific articles, including articles on which the CME questions are based, published in 2 anesthesiology journals Monday through Friday with a reminder to take the same test every six months; and group 3 will get e-mailed web links to blogs Monday through Friday based on the same specific articles as in group 2; each daily blog will focus on a specific article, including articles on which CME questions are based, the blogs will have web links to the articles on which they are based and every six months group 3 will get a reminder to take the same test. This will continue for 2 years' duration. Every six months, the investigators will assess knowledge of material contained in the two journals using CME material from the journals.

The investigators hypothesize that those participants randomized to group 3, the group that will receive web links to blogs, will stay more informed, as measured by the test score of CME-based questions. The investigators expect that both groups 1, usual care, and 2, e-mailed links to articles, will have a similar low score as the investigators found in a preliminary study of anesthesiologists who were presented with a set of journal-based CME questions.

Public Health Significance. This study will demonstrate the utility of journal based blogs as a support to physicians in their effort to remain up to date with developing medical knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Member of the American Society of Anesthesiologists (ASA)
* Must have granted ASA permission to receive email requests

Exclusion Criteria:

* Unwillingness to participate in the study
* Inability to read or write
* Younger than 26 years of age

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
CME testing | 2 years
  CME testing scores based on CME tests from 2 different anesthesiology journals

CONTACTS AND LOCATIONS:
Overall Officials: Lance Lichtor, M.D., Principal Investigator — Yale University

REFERENCES:
- [Background] Ende J. Learning about learning. J Gen Intern Med. 1995 Mar;10(3):172-3. doi: 10.1007/BF02599678. No abstract available. PMID 7769477
- [Background] Weil E, Tu JV. Quality of congestive heart failure treatment at a Canadian teaching hospital. CMAJ. 2001 Aug 7;165(3):284-7. PMID 11517643
- [Background] Antonelli Incalzi R, Pedone C, Pahor M, Onder G, Carbonin PU; Gruppo Italiano di Farmacovigilanza nell'Anziano. Trends in prescribing ACE-inhibitors for congestive heart failure in elderly people. Aging Clin Exp Res. 2002 Dec;14(6):516-21. doi: 10.1007/BF03327353. PMID 12674493
- [Background] Koczka CP, Geraldino-Pardilla LB, Goodman AJ, Gress FG. A nationwide survey of gastroenterologists and their acquisition of knowledge. Am J Gastroenterol. 2013 Jul;108(7):1033-5. doi: 10.1038/ajg.2012.309. PMID 23820990
- [Background] White JA, Anderson P. Learning by internal medicine residents: differences and similarities of perceptions by residents and faculty. J Gen Intern Med. 1995 Mar;10(3):126-32. doi: 10.1007/BF02599665. PMID 7769468
- [Background] Schein M, Paladugu R, Sutija VG, Wise L. What American surgeons read: a survey of a thousand Fellows of the American College of Surgeons. Curr Surg. 2000 May 1;57(3):252-258. doi: 10.1016/s0149-7944(00)00177-x. PMID 10930623
- [Background] Ahmadi-Abhari S, Soltani A, Hosseinpanah F. Knowledge and attitudes of trainee physicians regarding evidence-based medicine: a questionnaire survey in Tehran, Iran. J Eval Clin Pract. 2008 Oct;14(5):775-9. doi: 10.1111/j.1365-2753.2008.01073.x. PMID 19018910
- [Background] Nylenna M, Aasland OG. Doctors' learning habits: CME activities among Norwegian physicians over the last decade. BMC Med Educ. 2007 May 8;7:10. doi: 10.1186/1472-6920-7-10. PMID 17488507
- [Background] Kitchin DR, Applegate KE. Learning radiology a survey investigating radiology resident use of textbooks, journals, and the internet. Acad Radiol. 2007 Sep;14(9):1113-20. doi: 10.1016/j.acra.2007.06.002. PMID 17707320
- [Background] Lai CJ, Aagaard E, Brandenburg S, Nadkarni M, Wei HG, Baron R. Brief report: Multiprogram evaluation of reading habits of primary care internal medicine residents on ambulatory rotations. J Gen Intern Med. 2006 May;21(5):486-9. doi: 10.1111/j.1525-1497.2006.00432.x. PMID 16704393
- [Background] Hinkson CR, Kaur N, Sipes MW, Pierson DJ. Impact of offering continuing respiratory care education credit hours on staff participation in a respiratory care journal club. Respir Care. 2011 Mar;56(3):303-5. doi: 10.4187/respcare.00952. Epub 2010 Nov 16. PMID 21235846
- [Background] Bero L, Rennie D. The Cochrane Collaboration. Preparing, maintaining, and disseminating systematic reviews of the effects of health care. JAMA. 1995 Dec 27;274(24):1935-8. doi: 10.1001/jama.274.24.1935. No abstract available. PMID 8568988
- [Background] Antman EM, Lau J, Kupelnick B, Mosteller F, Chalmers TC. A comparison of results of meta-analyses of randomized control trials and recommendations of clinical experts. Treatments for myocardial infarction. JAMA. 1992 Jul 8;268(2):240-8. PMID 1535110
- [Background] Straus S, Haynes RB. Managing evidence-based knowledge: the need for reliable, relevant and readable resources. CMAJ. 2009 Apr 28;180(9):942-5. doi: 10.1503/cmaj.081697. No abstract available. PMID 19398741
- [Background] Weingart SD, Faust JS. Future evolution of traditional journals and social media medical education. Emerg Med Australas. 2014 Feb;26(1):62-6. doi: 10.1111/1742-6723.12192. No abstract available. PMID 24495063
- [Background] Cadogan M, Thoma B, Chan TM, Lin M. Free Open Access Meducation (FOAM): the rise of emergency medicine and critical care blogs and podcasts (2002-2013). Emerg Med J. 2014 Oct;31(e1):e76-7. doi: 10.1136/emermed-2013-203502. Epub 2014 Feb 19. PMID 24554447
- [Background] Bednarczyk J, Pauls M, Fridfinnson J, Weldon E. Characteristics of evidence-based medicine training in Royal College of Physicians and Surgeons of Canada emergency medicine residencies - a national survey of program directors. BMC Med Educ. 2014 Mar 21;14:57. doi: 10.1186/1472-6920-14-57. PMID 24650317
- [Background] Cook DA, Dupras DM, Thompson WG, Pankratz VS. Web-based learning in residents' continuity clinics: a randomized, controlled trial. Acad Med. 2005 Jan;80(1):90-7. doi: 10.1097/00001888-200501000-00022. PMID 15618102
- [Background] Wang AT, Sandhu NP, Wittich CM, Mandrekar JN, Beckman TJ. Using social media to improve continuing medical education: a survey of course participants. Mayo Clin Proc. 2012 Dec;87(12):1162-70. doi: 10.1016/j.mayocp.2012.07.024. Epub 2012 Nov 7. PMID 23141117
- [Background] Pitkin RM, Branagan MA, Burmeister LF. Accuracy of data in abstracts of published research articles. JAMA. 1999 Mar 24-31;281(12):1110-1. doi: 10.1001/jama.281.12.1110. PMID 10188662
- [Background] Pitkin RM, Branagan MA. Can the accuracy of abstracts be improved by providing specific instructions? A randomized controlled trial. JAMA. 1998 Jul 15;280(3):267-9. doi: 10.1001/jama.280.3.267. PMID 9676677
- [Background] Peacock PJ, Peters TJ, Peacock JL. How well do structured abstracts reflect the articles they summarize? European Science Editing. 2009;35(1):3-5. Accessed 26 November 2014
- [Background] Marcelo A, Gavino A, Isip-Tan IT, Apostol-Nicodemus L, Mesa-Gaerlan FJ, Firaza PN, Faustorilla JF Jr, Callaghan FM, Fontelo P. A comparison of the accuracy of clinical decisions based on full-text articles and on journal abstracts alone: a study among residents in a tertiary care hospital. Evid Based Med. 2013 Apr;18(2):48-53. doi: 10.1136/eb-2012-100537. Epub 2012 Jul 10. PMID 22782923
- [Background] Kristof N. Professors , we need you! International New York Times. February 17 2014
- [Background] Linzer M, Brown JT, Frazier LM, DeLong ER, Siegel WC. Impact of a medical journal club on house-staff reading habits, knowledge, and critical appraisal skills. A randomized control trial. JAMA. 1988 Nov 4;260(17):2537-41. PMID 3050179
- [Background] Kerfoot BP, DeWolf WC, Masser BA, Church PA, Federman DD. Spaced education improves the retention of clinical knowledge by medical students: a randomised controlled trial. Med Educ. 2007 Jan;41(1):23-31. doi: 10.1111/j.1365-2929.2006.02644.x. PMID 17209889
- [Background] Davis N, Davis D, Bloch R. Continuing medical education: AMEE Education Guide No 35. Med Teach. 2008;30(7):652-66. doi: 10.1080/01421590802108323. PMID 18777424
- [Background] Mills P, Timmis A, Huber K, Ector H, Lancellotti P, Masic I, Ivanusa M, Antoniades L, Aschermann M, Videvaek J, Laucevicius A, Mustonen P, Artigou JY, Vardas P, Stefanadis C, Chiariello M, Bolognese L, Ambrosio G, van der Wall EE, Kulakowski P, Pinto FJ, Apetrei E, Oganov RG, Kamensky G, Luscher TF, Lerch R, Haouala H, Sansoy V, Shumakov V, Tajer CD, Lau CP, Marquez M, Krittayaphong R, Arai K, Alfonso F; European Society of Cardiology (ESC) National Society Cardiovascular Journals Editors and ESC Affiliated Societies Cardiovascular Journals Editors. The role of European national journals in education. Rev Esp Cardiol. 2009 Dec;62(12):1494-7. doi: 10.1016/s1885-5857(09)73548-0. No abstract available. PMID 20038420
- [Background] Baethge C, Marx C, Griebenow R, Leuschner H. CME in a general medical journal: three-year evaluation of CME in Deutsches Arzteblatt. Teach Learn Med. 2010 Jul;22(3):229-32. doi: 10.1080/10401334.2010.488486. PMID 20563947
- [Background] Beynat J, Ben Mehidi A, Aubert JP, Bron AM, Massin P, Creuzot-Garcher C. RETIDIAB(R): assessment of a continuing medical education website for the improvement of diabetic retinopathy management. Diabetes Metab. 2011 Apr;37(2):118-23. doi: 10.1016/j.diabet.2010.08.009. Epub 2010 Dec 9. PMID 21145772
- [Background] Haynes RB. Of studies, syntheses, synopses, and systems: the "4S" evolution of services for finding current best evidence. ACP J Club. 2001 Mar-Apr;134(2):A11-3. No abstract available. PMID 11280129
- [Background] Mukohara K, Schwartz MD. Electronic delivery of research summaries for academic generalist doctors: a randomised trial of an educational intervention. Med Educ. 2005 Apr;39(4):402-9. doi: 10.1111/j.1365-2929.2005.02109.x. PMID 15813763
- [Background] Grad RM, Pluye P, Mercer J, Marlow B, Beauchamp ME, Shulha M, Johnson-Lafleur J, Wood-Dauphinee S. Impact of research-based synopses delivered as daily e-mail: a prospective observational study. J Am Med Inform Assoc. 2008 Mar-Apr;15(2):240-5. doi: 10.1197/jamia.M2563. Epub 2007 Dec 20. PMID 18096905
- [Background] Tanna GV, Sood MM, Schiff J, Schwartz D, Naimark DM. Do e-mail alerts of new research increase knowledge translation? A "Nephrology Now" randomized control trial. Acad Med. 2011 Jan;86(1):132-8. doi: 10.1097/ACM.0b013e3181ffe89e. PMID 21099399